Document Date: December 17, 2018

Statistical analysis: The prespecified primary behavioral endpoint was percent change across AHRS items after the five-day treatment conducted using a repeated-measures MANCOVA (rmMANCOVA) with group status as a between-subjects factor and time following randomization (one week and one month) and item (7 individual items) included as within-subject factors. In pre-specified analyses, only baseline AHRS score was used as a covariate. However, higher chlorpromazine equivalents (CPZE) 1 correlated significantly with higher baseline AHRS total (r=0.22, p=0.04) and PANSS P3 (r=0.30, p=0.005) scores, justifying its inclusion as an additional covariate for all analysis. Neither baseline AHRS or CPZE differed significantly between groups.

1. Woods SW. Chlorpromazine equivalent doses for the newer atypical antipsychotics. *J Clin Psychiatry* 2003; **64**(6): 663-7.